CLINICAL TRIAL: NCT06074939
Title: Building the Case for Action: A Situational Analysis to Guide the Implementation of Preventive Interventions in Adolescent Tobacco Use and Air Pollution Exposure
Brief Title: FRESHAIR4Life: Building the Case for Action
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Maastricht University (Other); University of York (Other); University of Edinburgh (Other); The Initiative (Unknown); Lungs Europe (Unknown); International Primary Care Respiratory Group (Unknown); University of Groningen (Other); University of Crete (Other); Ministry of Health, Kyrgyzstan (Other Government); Romanian Center for Studies in Family Medicine (Unknown); Makerere University (Other)
Responsible Party: Principal Investigator, Rianne MJJ van der Kleij, PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: 23-3075; 101095461 (Other Grant/Funding Number: Horizon Europe); 10063681; 10060974; 1006440 (Other Grant/Funding Number: UKRI)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use; Pollution; Exposure; Non-communicable Disease
Keywords: Implementation studies; Mixed-methods; Participatory research
MeSH Terms: conditions — Tobacco Use; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to understand the burden and determinants of tobacco use and air pollution (AP) exposure among mid- to late adolescents in Greece, the Kyrgyz Republic, Pakistan, Romania, and Uganda. This context-specific knowledge will be crucial for selecting, adapting, and implementing preventive interventions in the next phase of the project.

The main questions the investigators aim to answer are:

* What is the perceived burden of tobacco use and AP exposure among adolescents?
* What are the contextual drivers and behavioral determinants contributing to (prevention of) these risk factors?
* How do the dynamics between stakeholders influence prevention efforts?

In this study, data will be collected through interviews, focus group discussions, photovoice, document analysis, observations, personal exposure monitoring, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents: mid- to late-adolescents (14 to 21 years) within the target population;
* Family members: relatives in the first or second degree of (not necessarily participating) adolescents;
* Providers: any relevant stakeholder that is connected to adolescents through profession (e.g. school teacher, youth worker) and/or providers of (public) healthcare;
* Stakeholders: any relevant stakeholder with either a specific expertise, in-depth knowledge or overall overview on the subject, and in direct contact with the community (e.g. community member/leader, policy maker). Due to the community- and individual-level focus of this research, individuals associated with the tobacco industry are deliberately not included as stakeholders.

Exclusion Criteria:

- People living outside the target area or not in direct contact with the target population.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be performed in Greece, Romania, the Kyrgyz Republic, Pakistan and Uganda. These countries all have a high NCD burden but differ largely in contextual factors like population size (from 6.7 million in the Kyrgyz Republic to 231 million in Pakistan), population age (median age of 15.9 years in Uganda, up to 44.7 years in Greece), income classification (low in Uganda, low-middle in Pakistan and the Kyrgyz Republic, and high in Greece and Romania) and life expectancy (62.9 years in Uganda to 81.1 years in Greece).
  All countries will have an urban area as starting point (for logistical reasons and due to high prevalence of the vast majority of risk factors in urban areas), with either a peri-urban or rural community as second investigation site. Genders will equally be included in the situational analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Quantitative and qualitative evaluation of perceived clinical symptoms due to tobacco use and/or AP exposure | 1 day
Quantitative and qualitative evaluation and exploration of perceived psychological impact due to tobacco use and/or AP exposure | 1 day
Quantitative and qualitative evaluation and exploration of social factors relating to tobacco use and/or AP exposure | 1 day
Quantitative evaluation of the burden due to tobacco use and/or AP exposure by monitoring personal exposure to air borne particulates (PM 10, PM 2.5 and PM 1), temperature and relative humidity, using personal exposure (PE) monitors | 1 day
Qualitative evaluation and exploration of contextual drivers relevant to intervention implementation for prevention of tobacco and/or AP exposure, e.g. current strategies, local infrastructure and accessibility of resources. | 1 day
Qualitative evaluation and exploration of contextual drivers relevant to intervention implementation for prevention of tobacco and/or AP exposure, e.g. the influence of social media. | 1 day
Qualitative evaluation and exploration of contextual drivers relevant to intervention implementation for prevention of tobacco and/or AP exposure, e.g. the local socio-political climate, policy regulations and industry tactics. | 1 day
Qualitative evaluation and exploration of the relationship, power dynamics and (medical) hierarchies between adolescents, providers and other stakeholders. | 1 day
Quantitative and qualitative evaluation and exploration of determinants of behavior change in adolescents and providers relating to intervention implementation for prevention of tobacco and/or AP exposure. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Rianne MJJ van der Kleij, PhD, Principal Investigator — Leiden University Medical Center